CLINICAL TRIAL: NCT01972568
Title: A Phase IIb, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Multidose, 24-Week Study to Evaluate the Efficacy and Safety of Atacicept in Subjects With Systemic Lupus Erythematosus (SLE)
Brief Title: Efficacy and Safety of Atacicept in Systemic Lupus Erythematosus
Acronym: ADDRESS II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 700461-023; 2013-002773-21 (EudraCT Number)
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Results first posted 2017-10-26 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Atacicept; Placebo
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — TACI receptor-IgG Fc fragment fusion protein

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Atacicept 75 mg (Experimental)
  Interventions: Drug: Atacicept 75 milligram (mg)
- Atacicept 150 mg (Experimental)
  Interventions: Drug: Atacicept 150 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atacicept 75 milligram (mg) — Atacicept 75 mg will be administered as subcutaneous injection once weekly for 24 weeks.
  Arms: Atacicept 75 mg
Drug: Atacicept 150 mg — Atacicept 150 mg will be administered as subcutaneous injection once weekly for 24 weeks.
  Arms: Atacicept 150 mg
Drug: Placebo — Placebo matched to atacicept will be administered as subcutaneous injection once weekly for 24 weeks.
  Arms: Placebo

SUMMARY:
This is a multi-center, double-blind, randomized, Phase 2b trial to evaluate the efficacy of atacicept in subjects with systemic lupus erythematosus (SLE).

ELIGIBILITY:
Inclusion Criteria:

* Eligible male and female subjects, aged 18 years or older
* Must have at least moderately active SLE, as defined as SLE Disease Activity Index-2000 (SLEDAI-2K) score greater than or equal to [>=] 6 at screening visit
* At least 4 of the 11 American college of rheumatology (ACR) classification criteria for SLE (diagnosed >= 6 months prior to the screening visit)
* Be seropositive for anti-nuclear antibodies (ANA) and/or anti-double-stranded deoxyribonucleic acid (anti-dsDNA) antibodies
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Subjects have demyelinating disorder
* Severe central nervous system SLE
* Use of cyclophosphamide within 3 months of the screening visit
* Urine protein:creatinine ratio (UPCr) >= 2 milligram per milligram (mg/mg) per day
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono, Inc., Rockland MA, a subsidiary of Merck KGaA, Darmstadt, Germany
Locations (138):
- United States (30):
  - Pinnacle Research Group LLC, Anniston, Alabama
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - University of Alabama at Birmingham - (UAB), Birmingham, Alabama
  - Southern California Permanente Medical Group, Anaheim, California
  - Wallace Rheumatic Study Center, Los Angeles, California
  - East Bay Rheumatology Medical Group, Inc., San Leandro, California
  - Clinical Research of West Florida - Corporate, Dunedin, Florida
  - Center for Rheumatology, Immunology & Arthritis, Fort Lauderdale, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Goldpoint Clinical Research, LLC, Indianapolis, Indiana
  - AA MRC LLC Ahmed Arif Medical Research Center, Grand Blanc, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - North MS Medical Clinics, Inc., Tupelo, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - The Feinstein Institute for Medical Research, Manhasset, New York
  - Hospital for Special Surgery, New York, New York
  - Box Arthritis & Rheumatology of the Carolinas PLLC, Charlotte, North Carolina
  - MetroHealth System, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - STAT Research, Inc., Dayton, Ohio
  - Arthritis & Rheumatology Center of Oklahoma, Oklahoma City, Oklahoma
  - OMRF, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Clinical Research Center of Reading LLC, Wyomissing, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - UTMB Pathology Clinical Services, Galveston, Texas
  - Arthritis & Osteoporosis Clinic, Waco, Texas
  - Danville Orthopedic Clinic, Inc., Danville, Virginia
- Argentina (11):
  - APRILLUS, Ciudad Autonoma Buenos Aires
  - Atencion Integral en Reumatologia (AIR), Ciudad Autonoma Buenos Aires
  - Hospital Italiano, Ciudad Autonoma Buenos Aires
  - Organizacion Medica de Investigacion (OMI), Ciudad Autonoma Buenos Aires
  - Policlìnica Red Omip S.A - Ensayos Clinicos GC, Mar del Plata
  - Centro de Investigacion Pergamino SA, Pergamino
  - Cordis S.A., Salta
  - Centro Polivalente de Asistencia e Inv. Clinica CER, San Juan
  - Centro Integral de Reumatologia, San Miguel de Tucumán
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán
  - Investigaciones Clinicas Tucuman, San Miguel de Tucumán
- Brazil (4):
  - CPD - Centro de Pesquisas em Diabetes, Porto Alegre
  - CLION - Clínica de Oncologia da Bahia, Salvador
  - Clínica de Neoplasias Litoral Ltda., Santa Catarina
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto
- Bulgaria (6):
  - MHAT "Eurohospital" - Plovdiv, OOD, Plovdiv
  - Medical Center "Teodora", EOOD, Rousse
  - DCC "Sveta Anna", EOOD, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
  - Medical Center "Nov Rehabilitatsionen Tsentar", EOOD, Stara Zagora
  - MHAT-Targovishte, AD, Targovishte
- Chile (5):
  - Biomedica, Santiago
  - Centro de Estudios Reumatologicos, Santiago
  - Centro Medico Prosalud, Santiago
  - SOMEAL, Santiago
  - CINVEC - Centro de Investigacion Clinica V Region, Viña del Mar
- Czechia (4):
  - A-Shine, s.r.o., Pilsen
  - Revmatologicky Ustav, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - MEDICAL PLUS s.r.o., Uherské Hradiště
- Germany (7):
  - Kerckhoff-Klinik gGmbH, Bad Nauheim
  - Charite Universitaetsmedizin Berlin - Campus Charite Mitte, Berlin
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Rheumazentrum Ruhrgebiet, Herne
  - Universitaetsklinikum Schleswig-Holstein - Campus Kiel, Kiel
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz
- Italy (6):
  - Azienda Ospedaliero-Universitaria Consorziale Pol. di Bari, Bari
  - Presidio Ospedaliero Vittorio Emanuele, Catania
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Azienda Ospedaliero Universitaria San Martino, Genova
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia
- Japan (13):
  - St. Luke's International Hospital, Chūōku
  - NHO Kyushu Medical Center, Fukuoka
  - Toho University Ohashi Medical Center, Meguro-ku
  - Okayama University Hospital, Okayama
  - Kitasato University Hospital, Sagamihara-shi
  - Hokkaido University Hospital, Sapporo
  - Sapporo City General Hospital, Sapporo
  - Hakujujikai Sasebochuo Hospital, Sasebo-shi
  - Tohoku University Hospital, Sendai
  - Jichi Medical University Hospital, Shimotsuke-shi
  - National Center for Global Health and Medicine Hospital, Shinjuku
  - Yuaikai Tomishiro Chuo Hospital, Tomigusuku-shi
  - Tsukuba University Hospital, Tsukuba
- Mexico (10):
  - Investigacion y Biomedicina de Chihuahua, S.C., Chihuahua City
  - Icle S.C., Guadalajara
  - Unidad de Investigacion en Enfermedades Cronico Degenerativas SC, Guadalajara
  - Investigacion Clinica de Leon S.C., León
  - Morales Vargas Centro de Investigacion, S.C., León
  - Centro de Estudios Clinicos Especializados, Mérida
  - Accelerium S. de R.L. de C.V., Monterrey
  - ALIVIA Clínica de Alta Especialidad S.A. de C.V., Monterrey
  - Clinica de Enfermedades Cronicas y de Procedimientos Especiales, S.C., Morelia
  - Hospital Universitario de Saltillo "Dr. Gonzalo Valdés Valdés", Saltillo
- Peru (4):
  - Clinica El Golf, Lima
  - Clinica Medica Cayetano Heredia, Lima
  - Clinica Vesalio, Lima
  - HMA - Hospital Maria Auxiliadora, Lima
- Philippines (5):
  - Angeles University Foundation Medical Center, Angeles City
  - Mary Mediatrix Medical Center, Batangas
  - Davao Doctors Hospital, Davao City
  - Iloilo Doctors Hospital, Iloilo City
  - St. Luke's Medical Center, Quezon City
- Poland (4):
  - Szpital Uniwersytecki nr 2 im.dr J. Biziela, Bydgoszcz
  - Niepubliczny Zaklad Opieki Zdrowotnej "Nasz Lekarz" Praktyka Grupowa Lekarzy Rodzinnych z, Torun
  - Rheuma Medicus Zaklad Opieki Zdrowotnej, Warsaw
  - Wojskowy Instytut Medyczny, Warsaw
- Russia (11):
  - SBEI HPE Altai State Medical University of MoH and SD, Barnaul
  - SBHI of Kem. "Regional Clinical Hospital for War Veterans", Kemerovo
  - First Moscow State Medical University n.a. I.M. Sechenov, Moscow
  - Municipal City Hospital #2, Omsk
  - Republican Hospital n.a. V.A. Baranov, Petrozavodsk
  - Clinical Rheumatology Hospital #25, Saint Petersburg
  - Out - patient Clinic # 107, Saint Petersburg
  - City Clinical Hospital #12, Saratov
  - Regional Clinical Hospital, Saratov
  - Regional Clinical Hospital, Vladimir
  - Yaroslavl State Medical University, Yaroslavl
- South Africa (3):
  - Dr CE Spargo and Dr RB Bhorat, Cape Town
  - Naidoo, A, Durban
  - Winelands Medical Research Centre, Stellenbosch
- South Korea (5):
  - Gachon University Gil Medical Center, Incheon
  - Konkuk University Medical Center, Seoul
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Ajou University Hospital, Suwon
- Spain (4):
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital de Sagunto, Sagunto
  - Hospital Clínico Universitario de Valladolid, Valladolid
- United Kingdom (6):
  - Royal National Hospital for Rheumatic Diseases, Bath
  - Royal Sussex County Hospital, Brighton
  - University Hospital Coventry, Coventry
  - Guy's Hospital, London
  - University College London Hospitals, London
  - Wrightington Hospital, Wigan

REFERENCES:
- [Derived] Pitsiu M, Yalkinoglu O, Farrell C, Girard P, Vazquez-Mateo C, Papasouliotis O. Population pharmacokinetics of atacicept in systemic lupus erythematosus: An analysis of three clinical trials. CPT Pharmacometrics Syst Pharmacol. 2023 Aug;12(8):1157-1169. doi: 10.1002/psp4.12982. Epub 2023 Jun 18. PMID 37332136
- [Derived] Morand EF, Isenberg DA, Wallace DJ, Kao AH, Vazquez-Mateo C, Chang P, Pudota K, Aranow C, Merrill JT. Attainment of treat-to-target endpoints in SLE patients with high disease activity in the atacicept phase 2b ADDRESS II study. Rheumatology (Oxford). 2020 Oct 1;59(10):2930-2938. doi: 10.1093/rheumatology/keaa029. PMID 32107560
- [Derived] Merrill JT, Wallace DJ, Wax S, Kao A, Fraser PA, Chang P, Isenberg D; ADDRESS II Investigators. Efficacy and Safety of Atacicept in Patients With Systemic Lupus Erythematosus: Results of a Twenty-Four-Week, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Arm, Phase IIb Study. Arthritis Rheumatol. 2018 Feb;70(2):266-276. doi: 10.1002/art.40360. PMID 29073347

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 136 sites in 18 countries in Asia, Europe, North America, Central America, and South America.
Groups:
- Atacicept 75 mg: Subjects received atacicept 75 milligram (mg) as once-weekly subcutaneous injection for 24 weeks.
- Atacicept 150 mg: Subjects received atacicept 150 mg as once-weekly subcutaneous injection for 24 weeks.
- Placebo: Subjects received placebo matched to atacicept as once-weekly subcutaneous injection for 24 weeks.
Period: Overall Study
Arm/Group | Atacicept 75 mg | Atacicept 150 mg | Placebo
Started | 102 | 104 | 100
Completed | 86 | 92 | 84
Not Completed | 16 | 12 | 16
Not completed — Other events | 3 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 2
Not completed — Protocol Violation | 1 | 2 | 2
Not completed — Withdrawal by Subject | 6 | 3 | 7
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Adverse Event | 5 | 6 | 5

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) analysis set included all randomized subjects who had received at least 1 dose of investigational medicinal product (IMP).
Groups:
- Total: Total of all reporting groups
Arm/Group | Atacicept 75 mg | Atacicept 150 mg | Placebo | Total
Number analyzed (Participants) | 102 | 104 | 100 | 306
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (11.2) | 39 (11.6) | 40 (13.0) | 39 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 97 | 90 | 280
  Male | 9 | 7 | 10 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Systemic Lupus Erythematosus (SLE) Responder Index (SRI) Response at Week 24 Using Screening Visit as Baseline
Description: SRI response, a composite measure of reduced SLE disease activity, was defined as a reduction in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) disease activity score of greater than or equal to (>=) 4 points; no significant worsening in Physician's Global Assessment (PGA) score (<10 % increase, defined as <0.3 point increase for statistical analyses); no new British Isles Lupus Assessment Group (BILAG) A organ domain scores and <=1 (defined as no more than one) new BILAG B organ domain score.
Time Frame: Week 24
Population: mITT analysis set included all randomized subjects who had received at least 1 dose of IMP.
Measure: Number; unit: percentage of subjects
Arm/Group | Atacicept 75 mg | Atacicept 150 mg | Placebo
Number analyzed (Participants) | 102 | 104 | 100
percentage of subjects | 57.8 | 53.8 | 44.0
Statistical Analysis 1: Comparison: Atacicept 150 mg vs Placebo; Test type: Superiority or Other; p = 0.1208, Logistic regression model; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.89 to 2.72]

2. Secondary Outcome: Percentage of Subjects at Week 24 Whose Prednisone-Equivalent Corticosteroid (CS) Dose Reduced From Screening by >=25% and to a Dose of =<7.5mg/Day, and no British Isles Lupus Assessment Group (BILAG) A or 2B Flare in Disease Activity
Description: BILAG A or 2B flare is defined by 1 new BILAG A organ domain score and/or 2 new BILAG B organ domain scores compared to the Screening Visit. The BILAG disease activity index evaluates systemic lupus erythematosus (SLE) activity in 8 organ systems, using a separate alphabetic score (A to E) assigned to each organ system defined as follows. BILAG A: Disease sufficiently active requiring disease-modifying treatment (prednisone >20 mg daily or immunosuppressants); BILAG B: moderate disease activity requiring treatment with systemic low-dose oral glucocorticoids, intramuscular or intra-articular or soft tissue CS injection, topical CS or immunosuppressants, or symptomatic therapy such as antimalarials or NSAIDs. BILAG C: mild disease; BILAG D: system previously affected but now inactive and BILAG E: system never involved.
Time Frame: Week 24
Population: mITT analysis set included all randomized subjects who had received at least 1 dose of IMP. Here "Number of Participants Analyzed" signifies those subjects whose CS dose >=10 mg at Screening.
Measure: Number; unit: percentage of subjects
Arm/Group | Atacicept 75 mg | Atacicept 150 mg | Placebo
Number analyzed (Participants) | 56 | 53 | 53
percentage of subjects | 17.9 | 11.3 | 18.9

3. Secondary Outcome: Percentage of Subjects With Patient Global Impression of Change (PGIC) Categories at Week 24
Description: The PGIC is self-rated scale that asks the subject to describe the change in activity limitations, symptoms, emotions, and overall Quality of life (QoL) related to the subject's painful condition on the following scale: 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse) and 7 (very much worse). Percentage of subjects in the PGIC categories of very much or much improved (1 or 2), minimally improved or no change or minimally worse (3 or 4 or 5) and much or very much worse (6 or 7) at Week 24 were presented.
Time Frame: Week 24
Population: mITT analysis set included all randomized subjects who had received at least 1 dose of IMP.
Measure: Number; unit: percentage of subjects
Arm/Group | Atacicept 75 mg | Atacicept 150 mg | Placebo
Number analyzed (Participants) | 102 | 104 | 100
percentage of subjects
  Very much or much improved | 57.8 | 53.8 | 46.0
  Minimally improved or no change or minimally worse | 39.2 | 44.2 | 46.0
  Much or very much worse | 2.0 | 1.0 | 6.0
  Missing | 1.0 | 1.0 | 2.0

4. Secondary Outcome: Change From Screening in Prednisolone-Equivalent Corticosteroid (CS) Daily Dose at Week 24
Description: Change From screening visit to Week 24 of prednisolone-equivalent CS daily dose was presented.
Time Frame: Screening and Week 24
Population: mITT analysis set included all randomized subjects who had received at least 1 dose of IMP.
Measure: Mean (Standard Deviation); unit: mg per day
Arm/Group | Atacicept 75 mg | Atacicept 150 mg | Placebo
Number analyzed (Participants) | 102 | 104 | 100
mg per day | -2.64 (6.106) | -1.87 (4.653) | -1.89 (5.588)

5. Secondary Outcome: Time From Randomization to First SRI Response During Treatment Period
Description: SRI response, a composite measure of reduced SLE disease activity, was defined as a reduction in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) disease activity score of greater than or equal to (>=) 4 points; no significant worsening in Physician's Global Assessment (PGA) score (<10 % increase, defined as <0.3 point increase for statistical analyses); no new British Isles Lupus Assessment Group (BILAG) A organ domain scores and <=1 (defined as no more than one) new BILAG B organ domain score. Time to first SRI response during treatment period was presented.
Time Frame: Baseline up to 24 Weeks
Population: mITT analysis set included all randomized subjects who had received at least 1 dose of IMP.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Atacicept 75 mg | Atacicept 150 mg | Placebo
Number analyzed (Participants) | 102 | 104 | 100
weeks | 12.4 [12.1 to 16.7] | 16.1 [12.0 to 16.4] | 16.1 [12.1 to 20.1]

6. Secondary Outcome: Percentage of Subjects With British Isles Lupus Assessment Group (BILAG)-Based Combined Lupus Assessment (BICLA) Response at Week 24
Description: The BICLA response is defined as BILAG-2004 improvement (all screening visit BILAG A improving to B/C/D, all screening visit BILAG B to C/D, and <=1 new BILAG B and no new BILAG A); no deterioration in SLEDAI total score; PGA increase by <10% (defined as <0.3 point increase for the statistical analyses) and no nonpermitted medication/treatment.
Time Frame: Week 24
Population: mITT analysis set included all randomized subjects who had received at least 1 dose of IMP. Here "Number of Participants Analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Number; unit: percentage of subjects
Arm/Group | Atacicept 75 mg | Atacicept 150 mg | Placebo
Number analyzed (Participants) | 88 | 100 | 93
percentage of subjects | 53.4 | 49.0 | 45.2

7. Secondary Outcome: Percentage of Subjects With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An AE was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Treatment-emergent are events between first dose of study drug and up to 48 weeks. TEAEs include both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to 24 weeks after last dose of study drug (assessed up to maximum of 48 weeks)
Population: Safety analysis set included all randomized subjects who received at least 1 dose of IMP.
Measure: Number; unit: percentage of subjects
Arm/Group | Atacicept 75 mg | Atacicept 150 mg | Placebo
Number analyzed (Participants) | 102 | 104 | 100
percentage of subjects
  TEAEs | 81.4 | 80.8 | 72.0
  Serious TEAEs | 8.8 | 5.8 | 12.0

8. Secondary Outcome: Change From Week 0 (Day 1) in SF-36 Components at Week 24
Description: The 36-Item Short-Form Health Survey (SF-36) is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. These 8 aspects can also be summarized as physical and mental component summary scores. Total of 10 variables were analyzed (8 aspects, 2 component summary scores). The score for each of the 8 aspects and 2 component summary scores was scaled from 0 to 100, where 0 = lowest level of functioning and 100 = highest level of functioning.
Time Frame: Week 0 (Day 1) and Week 24
Population: mITT analysis set included all randomized subjects who had received at least 1 dose of IMP. Here "Number Analyzed" signifies those subjects who were evaluable for this outcome measure at specified categories.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atacicept 75 mg | Atacicept 150 mg | Placebo
Number analyzed (Participants) | 102 | 104 | 100
units on a scale
  Physical Component Summary: number analyzed (Participants) | 101 | 100 | 97
  Physical Component Summary | 4.7 (7.95) | 3.4 (7.57) | 3.5 (10.33)
  Mental Component Summary: number analyzed (Participants) | 101 | 100 | 97
  Mental Component Summary | 1.9 (12.01) | 1.8 (9.08) | 0.7 (11.44)
  Physical Functioning: number analyzed (Participants) | 85 | 89 | 82
  Physical Functioning | 3.5 (9.30) | 3.8 (8.42) | 3.3 (8.62)
  Role-Physical: number analyzed (Participants) | 85 | 89 | 82
  Role-Physical | 4.3 (10.26) | 2.3 (8.64) | 3.9 (9.51)
  Bodily Pain: number analyzed (Participants) | 85 | 89 | 82
  Bodily Pain | 6.0 (10.22) | 4.4 (9.30) | 5.6 (10.72)
  General Health: number analyzed (Participants) | 84 | 89 | 82
  General Health | 2.9 (8.43) | 3.0 (7.72) | 4.4 (8.00)
  Vitality: number analyzed (Participants) | 84 | 89 | 82
  Vitality | 3.9 (9.86) | 3.7 (9.76) | 3.5 (9.57)
  Social Functioning: number analyzed (Participants) | 85 | 89 | 82
  Social Functioning | 3.8 (11.45) | 2.2 (10.06) | 4.3 (11.08)
  Role-Emotional: number analyzed (Participants) | 85 | 89 | 82
  Role-Emotional | 2.5 (12.71) | 1.0 (10.43) | 2.3 (10.99)
  Mental Health: number analyzed (Participants) | 84 | 89 | 82
  Mental Health | 2.3 (12.30) | 2.8 (8.87) | 2.1 (10.60)

9. Post Hoc Outcome: High Disease Activity Subpopulation (SLEDAI-2K >=10 at Screening): Logistic Regression of Percentage of Subjects With SRI-6 Response at Week 24
Description: SRI-6 response, a composite measure of reduced SLE disease activity, was defined as a reduction in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) disease activity score of greater than or equal to (>=) 6 points; no significant worsening in Physician's Global Assessment (PGA) score (<10 % increase, defined as <0.3 point increase for statistical analyses); no new British Isles Lupus Assessment Group (BILAG) A organ domain scores and <=1 (defined as no more than one) new BILAG B organ domain score. Logistic regression of number of subjects with SRI-6 response was analyzed by using Logistic regression model.
Time Frame: Week 24
Population: mITT_HDA analysis set included mITT population with high disease activity (HDA) defined as screening SLE Disease Activity Index (SLEDAI) >=10.
Measure: Number; unit: percentage of subjects
Arm/Group | Atacicept 75 mg | Atacicept 150 mg | Placebo
Number analyzed (Participants) | 55 | 51 | 52
percentage of subjects | 43.6 | 54.9 | 28.8
Statistical Analysis 1: Comparison: Atacicept 150 mg vs Placebo; Test type: Superiority or Other; p = 0.0048, Logistic regression model; Odds Ratio (OR) = 3.31, 95% CI 2-sided [1.44 to 7.61]

10. Primary Outcome: Percentage of Subjects With Systemic Lupus Erythematosus (SLE) Responder Index (SRI) Response at Week 24 Using Day 1 as Baseline
Description: as for outcome 1
Time Frame: Week 24
Population: mITT analysis set included all randomized subjects who had received at least 1 dose of IMP.
Measure: Number; unit: percentage of subjects
Arm/Group | Atacicept 75 mg | Atacicept 150 mg | Placebo
Number analyzed (Participants) | 102 | 104 | 100
percentage of subjects | 55.9 | 55.8 | 41.0
Statistical Analysis 1: Comparison: Atacicept 150 mg vs Placebo; Test type: Superiority or Other; p = 0.0202, Logistic regression model; Odds Ratio (OR) = 1.96, 95% CI 2-sided [1.11 to 3.46]

ADVERSE EVENTS:
Time Frame: Baseline up to 24 weeks after last dose of study drug (assessed up to maximum of 48 weeks)
Arm/Group | Atacicept 75 mg | Atacicept 150 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 9/102 | 6/104 | 12/100
Other Adverse Events (participants affected / at risk) | 83/102 | 84/104 | 72/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atacicept 75 mg (N=102) | Atacicept 150 mg (N=104) | Placebo (N=100)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Mitral valve prolapse (Cardiac disorders) | 0 | 0 | 1
Right ventricular dilatation (Cardiac disorders) | 0 | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Abscess neck (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 1
Cardiac valve vegetation (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Endocarditis bacterial (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Infective aortitis (Infections and infestations) | 0 | 1 | 0
Lymph node abscess (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Ophthalmic herpes zoster (Infections and infestations) | 0 | 0 | 1
Parotitis (Infections and infestations) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Sinusitis bacterial (Infections and infestations) | 1 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Temporal lobe epilepsy (Nervous system disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atacicept 75 mg (N=102) | Atacicept 150 mg (N=104) | Placebo (N=100)
Diarrhoea (Gastrointestinal disorders) | 8 | 12 | 5
Nausea (Gastrointestinal disorders) | 9 | 5 | 1
Fatigue (General disorders) | 6 | 3 | 2
Injection site pain (General disorders) | 12 | 14 | 7
Injection site reaction (General disorders) | 42 | 43 | 19
Nasopharyngitis (Infections and infestations) | 6 | 7 | 5
Upper respiratory tract infection (Infections and infestations) | 10 | 13 | 3
Urinary tract infection (Infections and infestations) | 12 | 12 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 7
Headache (Nervous system disorders) | 11 | 15 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other